CLINICAL TRIAL: NCT01337401
Title: A Phase II Trial of Cediranib in the Treatment of Patients With Alveolar Soft Part Sarcoma (CASPS)
Brief Title: A Trial of Cediranib in the Treatment of Patients With Alveolar Soft Part Sarcoma (CASPS)
Acronym: CASPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICR-CTSU/2010/10027; 2010-021163-33 (EudraCT Number); CRUK/10/021 (Other Grant/Funding Number: Cancer Research UK); ISRCTN63733470 (Registry Identifier: Randomised controlled Trials); ISSRECE0036 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2011-04-11; First posted 2011-04-18 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Alveolar Soft-part Sarcoma
Keywords: Cediranib; ASPS; Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Sarcoma | interventions — cediranib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blinded Cediranib (Experimental)
  Interventions: Drug: Cediranib
- Blinded Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cediranib — 30mg once daily, oral until disease progression
  Arms: Blinded Cediranib
Drug: Placebo — 30mg, once daily, oral until 24 weeks or disease progression if sooner
  Arms: Blinded Placebo

SUMMARY:
The study is a two-arm, randomised, double-blind, international, multi-centre phase II trial of cediranib in Alveolar Soft Part Sarcoma (ASPS).

The study aims to confirm the ability of cediranib to halt disease progression in patients with metastatic ASPS, as measured by the change in tumour size at 24 weeks after randomisation, and to produce objective response according to RECIST criteria.

DETAILED DESCRIPTION:
Patients aged 16 years and older with a histologically confirmed diagnosis of ASPS will be recruited. Eligible patients will be randomised to receive cediranib (30 mg daily po) or placebo (30 mg daily po) in a 2:1 ratio. At 24 weeks post randomisation, treatment will be unblinded after which time all patients on placebo and those who have not progressed on active treatment will be given cediranib. Treatment will then continue until objective disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of ASPS (central confirmation not required at study entry)
2. Age 16 years and older
3. Availability of archived tissue blocks or unstained slides to enable confirmation of t(X;17) translocation
4. ECOG Performance Status of 0-1
5. Life expectancy of >12 weeks
6. Progressive disease as defined by RECIST v1.1 within 6 months prior to randomisation
7. Measurable metastatic disease using RECISTv1.1, i.e. at least one lesion 10 mm in diameter (15 mm in short axis for nodal lesions) assessable by CT (or MRI for brain metastases).
8. Patients with brain metastases are permitted provided disease is controlled with a stable dose of corticosteroid and/or non-enzyme inducing anticonvulsant
9. The capacity to understand the patient information sheet and ability to provide written informed consent
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
11. Able to swallow and retain oral medication

Exclusion Criteria:

1. Inadequate bone marrow reserve as demonstrated by an absolute neutrophil count ≤1.5 x 109/L or platelet count ≤100 x 109/L
2. Serum bilirubin ≥ 1.5 x ULN (unless Gilbert's syndrome)
3. ALT or AST ≥ 2.5 x ULN. If liver metastases are present, ALT or AST > 5 x ULN
4. Serum creatinine > 1.5 x ULN or a creatinine clearance (calculated or measured) of ≤ 50mL/min
5. Greater than +1 proteinuria unless urinary protein < 1.5g in a 24 hr period or protein/creatinine ratio < 1.5.
6. History of significant gastrointestinal impairment, as judged by the Investigator, that would significantly affect the absorption of cediranib.
7. Patients with a history of poorly controlled hypertension with resting blood pressure >150/100 mmHg in the presence or absence of a stable regimen of anti-hypertensive therapy.
8. Any evidence of severe or uncontrolled co-morbidities e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease, or active and uncontrolled infection.
9. Evidence of prolonged QTc >480 msec (using Bazetts correction, for which the formula is: QTc = QT/√RR) or history of familial long QT syndrome.
10. Significant recent haemorrhage (>30mL bleeding/episode in previous 3 months) or haemoptysis (>5mL fresh blood in previous 4 weeks).
11. Major thoracic or abdominal surgery in the 14 days prior to entry into the study, or a surgical incision that is not fully healed.
12. Pregnant or breast-feeding women; women of childbearing potential with a positive pregnancy test prior to receiving study medication; women the intention of pregnancy during study treatment; women of child bearing potential unwilling to have a urine or serum pregnancy test prior to study entry (even if surgically sterilised).
13. Men and women of childbearing potential unwilling to use adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilisation) for the duration of the study and should continue such precautions for 2 weeks after receiving the last study treatment.
14. History of anticancer (including investigational, non-registered) treatment in the four weeks prior to first dose of cediranib, with the exception of palliative radiotherapy for symptom control.
15. Previous treatment with cediranib.
16. Known hypersensitivity to any excipient of cediranib.
17. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within 5 years, unless the patient has been disease free for 2 years and there is a tissue diagnosis of the primary cancer of interest from a target lesion.
18. Other concomitant anti-cancer therapy (including LHRH agonists) except steroids
19. Recent history of thrombosis
20. Patients with brain metastases if they are symptomatic requiring increasing steroids in the previous six weeks to study entry or those with evidence of recent and/or active bleeding, or those causing uncontrolled seizures.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of cediranib in the treatment of ASPS by measuring the percentage change in the sum of target marker lesion diameters from randomisation to week 24 (or progression if sooner) compared to treatment with placebo. | 24 Weeks of treatment

SECONDARY OUTCOMES:
Response rate at week 24, best response using RECISTv1.1 and best reduction (%) in tumour size | 24 Weeks of treatment
Progression-free survival and percentage alive and progression-free at 12 months (APF12) | 12 months of treatment
Length of Overall survival | Patients will be followed up every 12 weeks
The safety and tolerability profile of cediranib in patients with ASPS | Assessments will be made at every study visit (8-12 weekly)

CONTACTS AND LOCATIONS:
Locations (11):
- Australia (2):
  - Princess Alexandra Hospital, Brisbane
  - Royal Prince Alfred Hospital, Sydney
- Spain (3):
  - Hospital Santa Cruz i Sant Pau, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (6):
  - Bristol Haematology and Oncology Centre, Bristol
  - Royal Marsden Hospital, London
  - University College London Hospital, London
  - Christie Hospital, Manchester
  - Royal Victoria Infirmary/Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals, Nottingham

REFERENCES:
- [Derived] Judson I, Morden JP, Kilburn L, Leahy M, Benson C, Bhadri V, Campbell-Hewson Q, Cubedo R, Dangoor A, Fox L, Hennig I, Jarman K, Joubert W, Kernaghan S, Lopez Pousa A, McNeil C, Seddon B, Snowdon C, Tattersall M, Toms C, Martinez Trufero J, Bliss JM. Cediranib in patients with alveolar soft-part sarcoma (CASPS): a double-blind, placebo-controlled, randomised, phase 2 trial. Lancet Oncol. 2019 Jul;20(7):1023-1034. doi: 10.1016/S1470-2045(19)30215-3. Epub 2019 May 31. PMID 31160249